CLINICAL TRIAL: NCT00587652
Title: A Prospective Trial of Methylene Blue Chromoendoscopy in Barrett's Esophagus
Brief Title: Methylene Blue Chromoendoscopy in Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Christopher J. Gostout MD, Mayo Clinic
Other Study IDs: 2114-02; IRUSEOMO164
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Barrett Esophagus
Keywords: Barrett Esophagus; Methylene blue; Chromoendoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Intermediate Segment Barrett's (2-4cm)
- 2: Long segment Barrett's (>4 cm)

SUMMARY:
This study is being done to:

Determine if a temporary dye applied to the esophagus identifies areas of dysplasia (pre-cancer). Determine if certain dye patterns indicate specific grades of dysplasia. Determine if overall endoscopy costs can be reduced with this dye technique. Determine if the dye could allow fewer biopsies to be obtained in the future.

DETAILED DESCRIPTION:
Although methylene blue has been used effectively to identify areas of SIM in several studies, its superiority in identifying dysplasia in the setting of Barrett's esophagus has been inconclusive. In all studies to date dysplastic yield was equivalent or better than protocol techniques while requiring fewer biopsies. Variations in study design, staining technique and inexperience in staining interpretation are some of the reasons. Our goal is to build on the techniques that have been shown to be effective, standardize them for the purposes of our study, and to objectively evaluate if MB directed biopsies are useful in screening Barrett's patients for dysplasia. At the time of EGD when length of Barrett's is determined, patients will be stratified into either intermediate (2-4cm) or long segment (>4cm) Barrett's. Short segment Barrett's esophagus patients will not be considered, as MB techniques have not proved beneficial in dysplasia detection as previously described 7.

ELIGIBILITY:
Inclusion Criteria:

* History of Barrett's with or without dysplasia
* Able to give consent

Exclusion Criteria:

* Pregnancy or women of child-bearing potential
* Active esophagitis
* Esophageal varices
* Esophageal cancer (history of or current)
* Hypersensitivity to methylene blue
* Severe renal impairment (creatinine>2.0)
* Known glucose-6-phosphate dehydrogenase (G-6-PD) deficiency
* Symptomatic coronary artery disease
* Coagulopathy (INR>/=1.5)
* Thrombocytopenia </= 20K/ul
* Previous esophageal ablative therapy (EMR,PDT, APC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for surveillance upper endoscopy to assess Barrett's esophagus.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Any dysplasia or adenocarcinoma detected over all biopsies using each method. | one year

SECONDARY OUTCOMES:
The association between staining patterns and histologic grade of the biopsies obtained using methylene blue will be assessed. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Gostout, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Rajan E, Burgart LJ, Gostout CJ. Endoscopic and histologic diagnosis of Barrett esophagus. Mayo Clin Proc. 2001 Feb;76(2):217-25. doi: 10.1016/S0025-6196(11)63133-9. PMID 11213314
- [Background] Gopal DV. Another look at Barrett's esophagus. Current thinking on screening and surveillance strategies. Postgrad Med. 2001 Sep;110(3):57-8, 61-2, 65-8. doi: 10.3810/pgm.2001.09.1018. PMID 11570206
- [Background] Canto MI, Setrakian S, Petras RE, Blades E, Chak A, Sivak MV Jr. Methylene blue selectively stains intestinal metaplasia in Barrett's esophagus. Gastrointest Endosc. 1996 Jul;44(1):1-7. doi: 10.1016/s0016-5107(96)70221-3. PMID 8836709
- [Background] Weston AP, Krmpotich PT, Cherian R, Dixon A, Topalosvki M. Prospective long-term endoscopic and histological follow-up of short segment Barrett's esophagus: comparison with traditional long segment Barrett's esophagus. Am J Gastroenterol. 1997 Mar;92(3):407-13. PMID 9068459
- [Background] Fennerty MB, Sampliner RE, McGee DL, Hixson LJ, Garewal HS. Intestinal metaplasia of the stomach: identification by a selective mucosal staining technique. Gastrointest Endosc. 1992 Nov-Dec;38(6):696-8. doi: 10.1016/s0016-5107(92)70567-7. No abstract available. PMID 1282115
- [Background] Canto MI. Vital staining and Barrett's esophagus. Gastrointest Endosc. 1999 Mar;49(3 Pt 2):S12-6. doi: 10.1016/s0016-5107(99)70518-3. No abstract available. PMID 10049441
- [Background] Canto MI, Setrakian S, Willis J, Chak A, Petras R, Powe NR, Sivak MV Jr. Methylene blue-directed biopsies improve detection of intestinal metaplasia and dysplasia in Barrett's esophagus. Gastrointest Endosc. 2000 May;51(5):560-8. doi: 10.1016/s0016-5107(00)70290-2. PMID 10805842
- [Background] Kiesslich R, Hahn M, Herrmann G, Jung M. Screening for specialized columnar epithelium with methylene blue: chromoendoscopy in patients with Barrett's esophagus and a normal control group. Gastrointest Endosc. 2001 Jan;53(1):47-52. doi: 10.1067/mge.2001.111041. PMID 11154488
- [Background] Sharma P, Topalovski M, Mayo MS, Weston AP. Methylene blue chromoendoscopy for detection of short-segment Barrett's esophagus. Gastrointest Endosc. 2001 Sep;54(3):289-93. doi: 10.1067/mge.2001.115728. PMID 11522967
- [Background] Canto MI, Yoshida T, Gossner L. Chromoscopy of intestinal metaplasia in Barrett's esophagus. Endoscopy. 2002 Apr;34(4):330-6. doi: 10.1055/s-2002-23640. No abstract available. PMID 11932792
- [Background] Canto MI. Methylene blue chromoendoscopy for Barrett's esophagus: coming soon to your GI unit? Gastrointest Endosc. 2001 Sep;54(3):403-9. doi: 10.1067/mge.2001.117958. No abstract available. PMID 11522995
- [Background] Wo JM, Ray MB, Mayfield-Stokes S, Al-Sabbagh G, Gebrail F, Slone SP, Wilson MA. Comparison of methylene blue-directed biopsies and conventional biopsies in the detection of intestinal metaplasia and dysplasia in Barrett's esophagus: a preliminary study. Gastrointest Endosc. 2001 Sep;54(3):294-301. doi: 10.1067/mge.2001.115732. PMID 11522968
- [Background] Tabuchi M, Sueoka N, Fujimori T. Videoendoscopy with vital double dye staining (crystal violet and methylene blue) for detection of a minute focus of early stage adenocarcinoma in Barrett's esophagus: a case report. Gastrointest Endosc. 2001 Sep;54(3):385-8. doi: 10.1067/mge.2001.116458. No abstract available. PMID 11522988
- [Background] Gangarosa LM, Halter S, Mertz H. Methylene blue staining and endoscopic ultrasound evaluation of Barrett's esophagus with low-grade dysplasia. Dig Dis Sci. 2000 Feb;45(2):225-9. doi: 10.1023/a:1005479619246. PMID 10711429
- [Background] Breyer HP, Silva De Barros SG, Maguilnik I, Edelweiss MI. Does methylene blue detect intestinal metaplasia in Barrett's esophagus? Gastrointest Endosc. 2003 Apr;57(4):505-9. doi: 10.1067/mge.2003.137. PMID 12665760
- [Background] Montgomery E, Bronner MP, Goldblum JR, Greenson JK, Haber MM, Hart J, Lamps LW, Lauwers GY, Lazenby AJ, Lewin DN, Robert ME, Toledano AY, Shyr Y, Washington K. Reproducibility of the diagnosis of dysplasia in Barrett esophagus: a reaffirmation. Hum Pathol. 2001 Apr;32(4):368-78. doi: 10.1053/hupa.2001.23510. PMID 11331953
- [Background] Katzka DA, Rustgi AK. Gastroesophageal reflux disease and Barrett's esophagus. Med Clin North Am. 2000 Sep;84(5):1137-61. doi: 10.1016/s0025-7125(05)70280-7. PMID 11026922
- [Background] Canto MI, Setrakian S, Willis JE, Chak A, Petras RE, Sivak MV. Methylene blue staining of dysplastic and nondysplastic Barrett's esophagus: an in vivo and ex vivo study. Endoscopy. 2001 May;33(5):391-400. doi: 10.1055/s-2001-14427. PMID 11396755
- [Background] Hackelsberger A, Gunther T, Schultze V, Manes G, Dominguez-Munoz JE, Roessner A, Malfertheiner P. Intestinal metaplasia at the gastro-oesophageal junction: Helicobacter pylori gastritis or gastro-oesophageal reflux disease? Gut. 1998 Jul;43(1):17-21. doi: 10.1136/gut.43.1.17. PMID 9771400
- [Background] Goldman AI. Issues in designing sequential stopping rules for monitoring side effects in clinical trials. Control Clin Trials. 1987 Dec;8(4):327-37. doi: 10.1016/0197-2456(87)90153-x. PMID 3327653
- [Background] Canto MI. Chromoendoscopy and magnifying endoscopy for Barrett's esophagus. Clin Gastroenterol Hepatol. 2005 Jul;3(7 Suppl 1):S12-5. doi: 10.1016/s1542-3565(05)00289-2. PMID 16012986